CLINICAL TRIAL: NCT01100801
Title: A Phase II Study of Genomic-guided 'Standard-of-care' Chemotherapy for in Advanced Gastric Cancer Patients
Brief Title: A Study of Genomic-guided 'Standard-of-care' Chemotherapy for in Advanced Gastric Cancer Patients
Acronym: 3G
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Cancer Centre, Singapore (Other); Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA01/01/10; 2010/00064 (Other: NHG Domain Specific Review Board)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Recurrent Gastric Cancer
Keywords: advanced; metastatic
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — titanium silicide; Cisplatin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TS-1 with cisplatin (Experimental): Chemotherapy injection (60mg/m2 cisplatin) will be given on day 1.
  14 days of Oral TS-1 (40mg/m²) will be prescribed. Subjects will take it after breakfast and evening meal on Day 1-14 of a 3-weekly treatment cycle. Each cycle is about 21 days.
  Interventions: Drug: TS-1 with cisplatin
- TS-1 with oxaliplatin (Experimental): Chemotherapy injection (100mg/m2 oxaliplatin) will be given on day 1.
  14 days of Oral TS-1 (40mg/m²) will be prescribed. Subjects will take it after breakfast and evening meal on Day 1-14 of a 3-weekly treatment cycle. Each cycle is about 21 days.
  Interventions: Drug: TS-1 with oxaliplatin

INTERVENTIONS:
Drug: TS-1 with cisplatin
  Other Names: TS-1 with cis-diamminedichloroplatinum
  Arms: TS-1 with cisplatin
Drug: TS-1 with oxaliplatin
  Other Names: TS-1 with 3rd-generation platinum analog
  Arms: TS-1 with oxaliplatin

SUMMARY:
This is an open, non-randomized, multicenter Phase II study evaluating cisplatin plus TS-1 or oxaliplatin plus TS-1 as first-line therapy in predicted 'responder' to platinum and fluoropyrimidine.

This study is planned in 3 centers in Singapore and Korea. A total of 30 subjects will be enrolled into each treatment arms. Each centers will recruit 15-25 subjects predicted to be 'responder' to platinum and fluoropyrimidine. The study will consist of a prescreening period, a screening period and a treatment period. A fresh tumour biopsy sample will be obtained during the prescreening period for gene expression profiling.

As this is a genomics guided trial, obtaining tissue biopsies is vital to the conduct of the trial.

Patients will have the primary in situ (requirement for entry into trial), endoscopic biopsy performed prior to 1st cycle.

DETAILED DESCRIPTION:
Gastric cancer is the world's second leading cause of cancer death. For patients with unresectable disease or recurrent disease after surgery, the main therapeutic option is chemotherapy. Chemotherapy can improve survival and quality of life in patients with advanced disease when compared with best supportive care alone.

Despite a large number of randomized trials, there is no consensus as to the best agent or regimen. In general, combination chemotherapy regimens provide higher response rates than do single agent, however, this translates into only a modest improvement in outcome with a trade off in increased treatment toxicities. The key challenge in managing patients with advanced gastric cancer is to identify the appropriate drugs for patients who might benefit for palliative chemotherapy.

Gastric cancer is a heterogeneous disease with differing chemosensitivities to anti-cancer drugs. Current selection of standard therapy is often empirical. Gene expression profiling has been shown to have the capability to dissect this heterogeneity allowing for sub-classification and risk-stratification of cancers according to their biological features and clinical outcome. Utilising gene expression data coupled with in-vitro, in-vivo or clinical response data is a promising strategy that may enable clinicians to match the right drug to the right patient.

The purpose of the study are:

1. Assess the feasibility of genomic-guided therapy
2. Evaluated treatment response of standard-of-care chemotherapy in an enriched patient groups defined as 'responder' based on genomic-guided therapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced, metastatic or recurrent gastric cancer for which convention therapy of a platinum/fluoropyrimidine combination is indicated
* Predicted 'responder' to platinum and fluoropyrimidine based on tumour expression signature derived from in-vitro sensitivity array
* At least one measurable defined by RECIST
* Age >=21 years old
* Performance status (ECOG) 0-2
* Life expectancy >3 months
* No significant problems for oral intake and drug administration
* Adequate organ functions:

bone marrow function (ANC = 1,500/uL, Platelet = 100,000/ uL, Hb = 8.0 g/dl) renal function: serum creatinine = UNL (if serum creatinine > ULN, creatinine clearance should be = 60 mL/min) hepatic function (Total bilirubin < 2 x UNL and AST/ALT levels < 3 x ULN without liver metastasis, total bilirubin < 3x ULN and AST/ALT levels < 5 x ULN with liver metastasis)

* Recovery from relevant toxicity to previous treatment before study entry
* Ability to understand and willingness to sign a written informed consent before study entry

Exclusion Criteria:

* Prior chemotherapy for gastric cancer except neoadjuvant or adjuvant systemic therapy if terminated at least 6 months before the start of treatment in this study
* Prior radiotherapy was administered to target lesions selected for this study
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
* Presence of symptomatic or progressing CNS metastasis
* Serious illness or medical conditions:

Congestive heart failure (NYHA class III or IV), unstable angina or myocardial infarction within the past 3 months Hepatic cirrhosis (= Child class B) Psychiatric disorder that may interfere with protocol compliance Active infection

* Known hypersensitivity to platinum or fluoropyrimidine.
* Pregnant or lactating woman. Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential
* Any patients judged by the investigator to be unfit to participate in the study
* Predicted 'non-responder' to platinum and fluoropyrimidine based on tumour expression signature derived from in- vitro sensitivity array

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Response Rate (RR) | 1 year
  To determine the response rate of cisplatin/TS-1 and oxaliplatin/TS-1 combination in predicted 'responders'

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Arai W, Hosoya Y, Hyodo M, Yokoyama T, Hirashima Y, Yasuda Y, Nagai H, Shirasaka T. Alternate-day oral therapy with TS-1 for advanced gastric cancer. Int J Clin Oncol. 2004 Jun;9(3):143-8. doi: 10.1007/s10147-004-0381-9. PMID 15221596
- [Background] Koizumi W. Chemotherapy for advanced gastric cancer: review of global and Japanese status. Gastrointest Cancer Res. 2007 Sep;1(5):197-203. PMID 19262709